CLINICAL TRIAL: NCT04715230
Title: Meth-OD: A Phase 2a Study of IXT-m200 in Patients With Toxicity From Methamphetamine Overdose
Brief Title: Meth-OD: A Study of IXT-m200 in Patients With Toxicity From Methamphetamine Overdose
Acronym: Meth-OD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on slower than anticipated enrollment leading to fund exhaustion.
Sponsor: InterveXion Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M200C-2101; U01DA053043 (NIH)
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-01

CONDITIONS: Methamphetamine Intoxication (Disorder)
MeSH Terms: interventions — Lorazepam; Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IXT-m200 (Experimental): IXT-m200 is a high-affinity chimeric anti-METH monoclonal antibody that is well-tolerated in healthy volunteers and in non-intoxicated people with METH use disorder. The total dose will be given over 10 min for the 0.5-g dose and over 20 min for the 1-, 1.5-, and 2-g doses.
  Interventions: Biological: IXT-m200
- Treatment as Usual (TAU) (Active Comparator): Lorazepam is a benzodiazepine that is safe and commonly used to treat agitation and dysphoria in the emergency setting. Haloperidol is commonly used to treat agitation due to psychosis.
  Interventions: Drug: Lorazepam; Drug: Haloperidol

INTERVENTIONS:
Biological: IXT-m200 — IXT-m200 binds METH with high selectivity and affinity. The product contains a murine METH-binding variable region and the constant domains of a human immunoglobulin G (IgG) 2κ. This antibody isotype was chosen because of the lower risk of immune response compared to an IgG1 or IgG3. IXT-m200 targets METH, does not rely on binding to any endogenous target for its action, and has been well-tolerated in previous clinical studies.
  Arms: IXT-m200
Drug: Lorazepam — Lorazepam is a benzodiazepine that is safe and commonly used to treat agitation and dysphoria in the emergency setting.
  Arms: Treatment as Usual (TAU)
Drug: Haloperidol — Haloperidol is commonly used to treat agitation due to psychosis.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The hypothesis of this multisite Phase 2a study is that IXT-m200 will be well-tolerated in patients with acute mild to moderate METH toxicity. A randomized, open label design will be used in which one dose of IXT-m200 will be compared to treatment-as-usual (TAU). Approximately 40 participants will be enrolled in 4 cohorts. A dose escalation approach will be used so that progressively higher IXT-m200 doses will be evaluated in each cohort. In conjunction with safety monitoring, this design assures the opportunity to observe early safety findings before any participants are exposed to the next higher dose. The randomization ratio for IXT-m200 versus TAU is defined as 4:1 for each cohort so that the number of participants receiving TAU equals the number receiving each dose of IXT-m200 at the end of the study.

Agitation scales and vital signs will be recorded to track effect of the antibody treatment versus TAU over time on agitation associated with METH use. While in the emergency department (ED), detailed and pertinent medical and psychiatric histories, and physical exam will be obtained, along with laboratory assessments and ECGs. In the ED, participants will give blood samples for analysis of METH and IXT-m200 concentrations and followed for development of adverse events. Participants will be evaluated at 2 days and 4 weeks after discharge from the ED for adverse events and drug use history. Cohort escalation reviews will be performed by the Sponsor, Medical Monitor, and Data and Safety Monitoring Board (DSMB) between cohorts and the next group will not start until after completion of this review.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 to 45 years, inclusive;
2. Present to the ED with METH toxicity as defined in protocol;
3. Have a PANSS-EC score of 14-28, inclusive;
4. Have or agrees to have an intravenous (IV) line placed;
5. Give a history of METH use in the past 24 hours, with participant or observer attribution of symptoms to METH, or have a positive METH drug screen;
6. Be accompanied or readily represented by a legally authorized representative (surrogate) who can consent to participation on behalf of the participant; and
7. Assent to participation in the study.

Exclusion Criteria:

1. Present with concomitant opioid overdose requiring ventilatory support;
2. Be self-reported to be pregnant or lactating;
3. Be considered to have significant concomitant medical illness or trauma, or symptoms of severe METH toxicity including

   1. sepsis or febrile illness;
   2. myocardial infarction, cardiac decompensation or arrhythmias including tachycardia that is not sinus; severe hypertension (>180/110 mmHg); inadequately treated hypertension on chronic medication; history of vasculitis
   3. coma, stroke or severe head injury; new or ongoing seizure activity
   4. acute pulmonary decompensation or severe chronic obstructive pulmonary disease;
   5. any hepatic impairment and/or acute hepatitis or renal impairment due to concomitant medical illness; or
   6. current, or history of, neuroleptic malignant syndrome
4. Be considered to be at imminent risk of suicide or have disqualifying answers to the following two questions. Disqualifying answers would be 1b2 or 2b. 1. In the past 30 days, have you considered killing yourself? a) No; b) Yes - if Yes, how often? b1) Not often (twice or less), b2) Somewhat often (more than twice). 2. In the past year, have you attempted to kill yourself? a) No; b) Yes;
5. Be considered to be at imminent risk of injury or danger to self, others or property;
6. Have a history of severe allergy (rash, hives, breathing difficulty, etc.), known hypersensitivity or infusion reaction to any antibody medications, lorazepam or haloperidol; or
7. Be judged by the treating ED physician, investigator, or Sponsor (or designee) to be inappropriate for the study, including people whom the investigator determines cannot reasonably be consulted for assent to participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — InterveXion Therapeutics
Locations (4):
- United States (4):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Providence Regional Medical Center Everett, Everett, Washington
  - Sacred Heart Medical Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Final datasets are expected to contain IXT-m200 and METH concentration data, ACES scores over time, and safety data. No individually identifiable private information will be distributes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: These datasets will be available for distribution following submission to the FDA of the Clinical Study Report and publication. They will be available for 2 years after the initial publication.
Access Criteria: These datasets and associated documentation will be made available on CD by the Sponsor to requestors under a data sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology and not distributing to third parties; and (3) a commitment to destroying or returning the data after analyses are completed. Requests should be sent to intervexion@gmail.com

RESULTS

PARTICIPANT FLOW:
Groups:
- IXT-m200 Low Dose (0.5 g): IXT-m200 is a high-affinity chimeric anti-METH monoclonal antibody that is well-tolerated in healthy volunteers and in non-intoxicated people with METH use disorder. The total dose will be given over 10 min for the 0.5-g dose.
  IXT-m200: IXT-m200 binds METH with high selectivity and affinity. The product contains a murine METH-binding variable region and the constant domains of a human immunoglobulin G (IgG) 2κ. This antibody isotype was chosen because of the lower risk of immune response compared to an IgG1 or IgG3. IXT-m200 targets METH, does not rely on binding to any endogenous target for its action, and has been well-tolerated in previous clinical studies.
- IXT-m200 High Dose (2 g): IXT-m200 is a high-affinity chimeric anti-METH monoclonal antibody that is well-tolerated in healthy volunteers and in non-intoxicated people with METH use disorder. The total dose will be given over 20 min for the 2-g doses.
  IXT-m200: IXT-m200 binds METH with high selectivity and affinity. The product contains a murine METH-binding variable region and the constant domains of a human immunoglobulin G (IgG) 2κ. This antibody isotype was chosen because of the lower risk of immune response compared to an IgG1 or IgG3. IXT-m200 targets METH, does not rely on binding to any endogenous target for its action, and has been well-tolerated in previous clinical studies.
Period: Overall Study
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Started | 8 | 8 | 4
Completed | 7 | 3 | 3
Not Completed | 1 | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 8 | 8 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (6.23) | 36.8 (6.48) | 35.3 (7.17) | 35.5 (6.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 0 | 6
  Male | 6 | 4 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 6 | 7 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 6 | 6 | 4 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-related Adverse Events (AEs) as Measured by Vital Signs
Description: Blood pressure, heart rate, and temperature
Time Frame: 28 days
Population: All participants receiving a dose of IXT-m200 or TAU.
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Patients With Treatment-related AEs as Measured by Physical Examinations
Description: Physical examinations
Time Frame: 28 days
Population: All participants receiving a dose of IXT-m200 or TAU
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Patients With Treatment-related AEs as Measured by Clinical Laboratory Testing
Description: Clinical laboratory testing
Time Frame: 3 days
Population: All participants receiving a dose of IXT-m200 or TAU.
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Patients With Treatment-related AEs as Measured by Electrocardiogram
Description: Electrocardiogram
Time Frame: 4 hours
Population: All participants receiving a dose of IXT-m200 or TAU.
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
Participants | 0 | 0 | 0

5. Secondary Outcome: Time Course and Degree of Normalization of Agitation
Description: Agitation/sedation scores over time as measured by Agitation/Calmness Evaluation Score (ACES). The minimum value is 1 (highly agitated) and the highest value is 9 (completely sedated). A score of 3-5 is considered normal.
Time Frame: Baseline and hours 0.5, 1, 2, 3, 4, and 8 post-dose or until discharge.
Population: All participants receiving a dose of IXT-m200 or TAU. No further data were collected after participants were discharged. Some time points do not contain results as all participants in that group had been discharged prior to that timepoint or all data were missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
score on a scale
  Baseline | 2.1 (0.64) | 2. (0.53) | 2.8 (0.50)
  0.5 hour | 4.1 (1.81) | 3.6 (1.60) | 3.9 (1.67)
  1 hour | 4.6 (1.92) | 3.9 (1.81) | 5.8 (1.89)
  2 hours: number analyzed (Participants) | 7 | 7 | 4
  2 hours | 4.0 (1.91) | 4.0 (2.08) | 4.8 (0.50)
  3 hours: number analyzed (Participants) | 1 | 2 | 0
  3 hours | 7.0 | 3.0 (2.83) |
  4 hours: number analyzed (Participants) | 0 | 1 | 0
  4 hours |  | 1.0 |

6. Secondary Outcome: Number of Participants at Certain Degrees of Normalization of Blood Pressure Over Time
Description: Blood pressure over time; reported as the number of participants with blood pressure out of normal range (i.e., diastolic >110 or <50 mmHg, or systolic >180 or <90 mmHg))
Time Frame: Baseline and hours 0.5, 1, 2, 3, 4, and 8 post-dose or until discharge.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
Participants
  Baseline: High | 0 | 2 | 0
  Baseline: Normal | 8 | 5 | 4
  Baseline: Low | 0 | 1 | 0
  0.5 hour: number analyzed (Participants) | 8 | 8 | 3
  0.5 hour: High | 0 | 1 | 0
  0.5 hour: Normal | 8 | 7 | 3
  0.5 hour: Low | 0 | 0 | 0
  1 hour: High | 0 | 1 | 0
  1 hour: Normal | 8 | 7 | 4
  1 hour: Low | 0 | 0 | 0
  2 hours: number analyzed (Participants) | 7 | 5 | 2
  2 hours: High | 0 | 0 | 0
  2 hours: Normal | 7 | 5 | 1
  2 hours: Low | 0 | 0 | 1
  3 hours: number analyzed (Participants) | 1 | 2 | 0
  3 hours: High | 0 | 0 |
  3 hours: Normal | 1 | 2 |
  3 hours: Low | 0 | 0 |
  Prior to discharge: number analyzed (Participants) | 0 | 1 | 1
  Prior to discharge: High |  | 1 | 0
  Prior to discharge: Normal |  | 0 | 1
  Prior to discharge: Low |  | 0 | 0

7. Secondary Outcome: Number of Participants at Certain Degrees of Normalization of Heart Rate Over Time
Description: Heart rate over time reported as number of participants with heart rate high (>120 beats/min), normal, or low (<40 beats/min).
Time Frame: Baseline and hours 0.5, 1, 2, 3, 4, and 8 post-dose or until discharge.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
Participants
  Baseline: High | 0 | 0 | 0
  Baseline: Normal | 8 | 8 | 4
  Baseline: Low | 0 | 0 | 0
  0.5 hour: number analyzed (Participants) | 8 | 8 | 3
  0.5 hour: High | 1 | 0 | 0
  0.5 hour: Normal | 7 | 8 | 3
  0.5 hour: Low | 0 | 0 | 0
  1 hour: High | 1 | 0 | 0
  1 hour: Normal | 7 | 8 | 4
  1 hour: Low | 0 | 0 | 0
  2 hours: number analyzed (Participants) | 7 | 5 | 2
  2 hours: High | 1 | 0 | 0
  2 hours: Normal | 6 | 5 | 2
  2 hours: Low | 0 | 0 | 0
  3 hours: number analyzed (Participants) | 1 | 2 | 0
  3 hours: High | 0 | 0 |
  3 hours: Normal | 1 | 2 |
  3 hours: Low | 0 | 0 |
  Prior to discharge: number analyzed (Participants) | 0 | 1 | 1
  Prior to discharge: High |  | 0 | 0
  Prior to discharge: Normal |  | 1 | 1
  Prior to discharge: Low |  | 0 | 0

8. Secondary Outcome: Time Course and Degree of Normalization of Temperature
Description: Temperature over time
Time Frame: Baseline and hours 0.5, 1, 2, 3, 4, and 8 post-dose or until discharge.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 6 | 6 | 4
degrees Fahrenheit
  Baseline | 98.2 (0.62) | 98.25 (0.345) | 98.10 (0.424)
  0.5 hour: number analyzed (Participants) | 2 | 5 | 0
  0.5 hour | 98.05 (0.495) | 98.52 (0.476) |
  1 hour: number analyzed (Participants) | 2 | 4 | 1
  1 hour | 98.45 (0.778) | 98.48 (0.562) | 97.7
  2 hours: number analyzed (Participants) | 2 | 4 | 1
  2 hours | 98.50 (1.414) | 98.38 (0.907) | 97.7
  3 hours: number analyzed (Participants) | 1 | 1 | 0
  3 hours | 99.10 | 99.50 |
  Discharge: number analyzed (Participants) | 2 | 1 | 1
  Discharge | 97.40 (0.141) | 98.0 | 98.10

9. Secondary Outcome: Number of Participants Requiring Rescue Medications for Psychiatric or Cardiovascular Manifestations of METH Toxicity
Description: Number of participants that need rescue medications to treat:
  * agitation, dysphoria, or psychosis (central nervous system toxicity)
  * hypertension, tachycardia, or other cardiovascular instability (cardiovascular toxicity)
Time Frame: 8 hours
Population: All participants receiving a dose of IXT-m200 or TAU.
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
Participants
  Required rescue medications | 0 | 0 | 0
  Did not require rescue medications | 8 | 8 | 4

10. Other Pre Specified Outcome: Length of Patient Stay in the ED
Description: ED length of stay as measured by discharge time minus start of treatment time
Time Frame: Start of treatment until discharge
Population: All participants receiving a dose of IXT-m200 or TAU.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 8 | 4
hours | 8.940 (5.6843) | 8.031 (6.0973) | 10.196 (8.0826)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | IXT-m200 Low Dose (0.5 g) | IXT-m200 High Dose (2 g) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 5/8 | 2/8 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IXT-m200 Low Dose (0.5 g) (N=8) | IXT-m200 High Dose (2 g) (N=8) | Treatment as Usual (TAU) (N=4)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0) — Orbital Mass
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) — Increased liver enzymes and ongoing bilirubin
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IXT-m200 Low Dose (0.5 g) (N=8) | IXT-m200 High Dose (2 g) (N=8) | Treatment as Usual (TAU) (N=4)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide Sponsor opportunity to review proposed publications/disclosures before submission/disclosure. The first publication is to be a joint publication involving all sites, with Sponsor in control of such publication. Afterward, and if such publication is not made within 12 months following finalization of the clinical study report or termination of the study at all sites, PI may publish separately.

DOCUMENTS (3):
  • Study Protocol (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT04715230/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT04715230/SAP_001.pdf
  • Informed Consent Form (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT04715230/ICF_002.pdf